CLINICAL TRIAL: NCT05246943
Title: The Correlation of a D-dimer Testing Protocol With Venous Thromboembolism in Surgical Colorectal Patients
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0266
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Venous Thromboses; Colorectal Cancer; Diverticular Diseases; Crohn Disease; Ulcerative Colitis; Deep Vein Thrombosis
Keywords: D-dimer; Colorectal Surgery; Thrombosis; DVT
MeSH Terms: conditions — Venous Thrombosis; Colorectal Neoplasms; Diverticular Diseases; Crohn Disease; Colitis, Ulcerative; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UTMB's Colorectal Surgical Cohort: Subjects who meet the inclusion criteria that will have colorectal surgery at UTMB
  Interventions: Diagnostic Test: D-dimer and lower limb venous duplex

INTERVENTIONS:
Diagnostic Test: D-dimer and lower limb venous duplex — D-dimer blood test- The D-dimer assay detects the presence of fibrin degradation products, which can indicate the breakdown of a fibrin clot Lower Limb Venous Duplex- Using an ultrasound to visually look for a clot

SUMMARY:
The purpose of this study is to evaluate the use of a D-dimer based protocol to screen for thrombotic events in colorectal surgical patients. This study is unique because of the multistage screening process for DVT's using a standardized D-dimer testing methodology and ultrasound that will take place throughout the preoperative, perioperative, and postoperative processes. The data collected from this screening study will help establish the baseline DVT rates in UTMB's colorectal surgical patients before and after surgery. Additionally, the data from this study can help determine if a D-dimer blood test has predictive value in UTMB's colorectal surgical patient population. This study may also provide preliminary evidence for further research regarding the adjustment of D-dimer cutoff values. Specifically for patient subsets such as surgical colorectal patients with a moderate pretest probability and clinical conditions associated with low test specificity

DETAILED DESCRIPTION:
This will be a quantitative prospective cohort study conducted at the University of Texas Medical Branch (UTMB) Galveston and League City campuses. Candidates include subjects who will have elective colorectal surgery at UTMB. This study looks to enroll 100 subjects who meet inclusion criteria. The subjects will undergo screening for DVT using a lower limb bilateral venous duplex and a plasma D-dimer assay no longer than 10 days before their operation. This data will be used to observe the point prevalence of DVT's in preoperative colorectal subjects prior to having colorectal surgery. On the day of surgery, the subject will have a D-dimer test. After the operation, for next 2 days the subjects will have a daily D-dimer test and a lower limb bilateral venous duplex on the second day only. This data will determine the incidence of DVT's that were detected by lower limb bilateral venous duplex on inpatient stay day 2 and possibly indicated by an upward trending D-dimer value during the first 2 days of the inpatient stay. Approximately 2 weeks after surgery, at the postoperative clinic appointment, the subject will have a D-dimer assay and a lower limb bilateral venous duplex. This information will be used to determine the number of DVT events in postoperative colorectal hospitalized subjects that were on the D-dimer monitoring protocol. The D-dimer assay detects the presence of fibrin degradation products, which may indicate a fibrin blood clot in the body.6 A maximum of 5 milliliters of blood will be collected for each D-dimer test. If a DVT is detected by the gold standard method which is a bilateral lower limb duplex during any point of study, the subject will be treated as per standard of care at UTMB by the colorectal surgical team

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer requiring surgical intervention-elective

   a)Benign or Malignant
2. Inflammatory colorectal conditions requiring surgical intervention-elective

   1. Diverticulitis
   2. Ulcerative Colitis
   3. Crohn's Disease

Exclusion Criteria:

* Pregnancy
* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a quantitative prospective cohort study conducted at the University of Texas Medical Branch (UTMB) Galveston and League City campuses. Candidates include subjects who will have elective colorectal surgery at UTMB.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Observe the point prevalence of DVT's in preoperative colorectal patients at UTMB prior to having colorectal surgery. | 1 year
  The data will be used to discover the prevalence of DVT prior to surgery and to establish DVT baseline rates at UTMB.
Determine the incidence of postoperative DVT that occurred during the first 2 days of the inpatient stay that was discovered by a lower limb venous duplex | 1 year
  Subjects will have a venous duplex on day two after surgery to look for a DVT
Compare the number of DVT events in postoperative hospitalized patients that were on the D-dimer monitoring protocol. | 1 year
  The data will be used to determine the number of DVT's that were discovered in the subject population and to establish baseline rates of DVT after surgery and hospital discharge
Determine if there is a statistical difference between the D-dimer value of patients with DVT prior to surgery compared to patients who develop DVT after surgery | 1 year
  This data will be used to compare the D-dimer values in subjects that had DVT prior to surgery to those who developed a postoperative DVT while inpatient or at the postoperative clinic appointment
Compare the D-dimer results of DVT positive subjects to DVT negative subjects to identify a specific result range seen in the DVT positive subjects. | 1 year
  These results will be used as preliminary evidence for future research to determine if revised D-dimer cut off values can be diagnostic in conditions known to have low test specificity

CONTACTS AND LOCATIONS:
Overall Officials: Uma Phatak, MD, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garg R, Mohammed A, Singh A, Regueiro M, Click B. Trends and Outcomes of Acute Diverticulitis in Inflammatory Bowel Disease: A Propensity-matched National Study. Inflamm Bowel Dis. 2022 Jan 5;28(1):48-53. doi: 10.1093/ibd/izab017. PMID 33528011
- [Result] Colorectal Writing Group for Surgical Care and Outcomes Assessment Program-Comparative Effectiveness Research Translation Network (SCOAP-CERTAIN) Collaborative; Nelson DW, Simianu VV, Bastawrous AL, Billingham RP, Fichera A, Florence MG, Johnson EK, Johnson MG, Thirlby RC, Flum DR, Steele SR. Thromboembolic Complications and Prophylaxis Patterns in Colorectal Surgery. JAMA Surg. 2015 Aug;150(8):712-20. doi: 10.1001/jamasurg.2015.1057. PMID 26060977
- [Result] Rees PA, Clouston HW, Duff S, Kirwan CC. Colorectal cancer and thrombosis. Int J Colorectal Dis. 2018 Jan;33(1):105-108. doi: 10.1007/s00384-017-2909-2. Epub 2017 Nov 10. PMID 29127473
- [Result] Stender MT, Frokjaer JB, Larsen TB, Lundbye-Christensen S, Thorlacius-Ussing O. Preoperative plasma D-dimer is a predictor of postoperative deep venous thrombosis in colorectal cancer patients: a clinical, prospective cohort study with one-year follow-up. Dis Colon Rectum. 2009 Mar;52(3):446-51. doi: 10.1007/DCR.0b013e318197e2b2. PMID 19333044
- [Result] Buchberg B, Masoomi H, Lusby K, Choi J, Barleben A, Magno C, Lane J, Nguyen N, Mills S, Stamos MJ. Incidence and risk factors of venous thromboembolism in colorectal surgery: does laparoscopy impart an advantage? Arch Surg. 2011 Jun;146(6):739-43. doi: 10.1001/archsurg.2011.127. PMID 21690452
- [Result] Johnson ED, Schell JC, Rodgers GM. The D-dimer assay. Am J Hematol. 2019 Jul;94(7):833-839. doi: 10.1002/ajh.25482. Epub 2019 Apr 19. PMID 30945756
- [Result] Weitz JI, Fredenburgh JC, Eikelboom JW. A Test in Context: D-Dimer. J Am Coll Cardiol. 2017 Nov 7;70(19):2411-2420. doi: 10.1016/j.jacc.2017.09.024. PMID 29096812
- [Result] Tassiopoulos AK, Mofakham S, Rubano JA, Labropoulos N, Bannazadeh M, Drakos P, Volteas P, Cleri NA, Alkadaa LN, Asencio AA, Oganov A, Hou W, Rutigliano DN, Singer AJ, Vosswinkel J, Talamini M, Mikell CB, Kaushansky K. D-Dimer-Driven Anticoagulation Reduces Mortality in Intubated COVID-19 Patients: A Cohort Study With a Propensity-Matched Analysis. Front Med (Lausanne). 2021 Feb 4;8:631335. doi: 10.3389/fmed.2021.631335. eCollection 2021. PMID 33634153
- [Result] Jiang Y, Li J, Liu Y, Zhang W. Diagnostic accuracy of deep vein thrombosis is increased by analysis using combined optimal cut-off values of postoperative plasma D-dimer levels. Exp Ther Med. 2016 May;11(5):1716-1720. doi: 10.3892/etm.2016.3125. Epub 2016 Mar 2. PMID 27168793